CLINICAL TRIAL: NCT00602836
Title: Phase II Trial of Pentostatin, Cyclophosphamide, and Rituximab Followed by Consolidation With Lenalidomide for Previously Untreated B-Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Rituximab, Pentostatin, Cyclophosphamide, and Lenalidomide in Treating Patients With Previously Untreated B-Cell Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582676; P30CA015083 (NIH); MC0784 (Other: Mayo Clinic Cancer Center); 07-002156 (Other: Mayo Clinic IRB); RV-CLL-PI-146 (Other: Celgene Protocol); NCI-2009-01281 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-01-12; First posted 2008-01-28 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2017-09

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; Lenalidomide; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PCR-Lenalidomide (Experimental): Pentostatin, Cyclophosphamide, Rituximab + Lenalidomide
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Lenalidomide; Drug: Pentostatin

INTERVENTIONS:
Biological: Rituximab — Cycle 1: 100 mg by IV on day 1, 375 mg/m^2 by IV on day 2 Cycle 2-6: 375 mg/m^2 by IV on day 1 (every 21 days)
Drug: Cyclophosphamide — 600 mg/m^2 by IV on day 1 of cycles 1-6 (every 21 days)
Drug: Lenalidomide — Cycle 7: 5 mg orally daily on days 1-28 Cycle 8: 10 mg orally daily on days 1-28 as tolerability permits Cycle 9 and beyond: 10 mg orally daily on days 1-28
Drug: Pentostatin — 2 mg/m^2 by IV on day 1 of cycles 1-6 (every 21 days)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as pentostatin and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Lenalidomide may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving rituximab together with combination chemotherapy and lenalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with pentostatin, cyclophosphamide, and lenalidomide works in treating patients with previously untreated B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the rate of complete and overall response using pentostatin, cyclophosphamide, and rituximab (PCR) followed by consolidation with lenalidomide in patients with previously untreated B-cell chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma.

Secondary

* To assess the proportion of patients who convert from a nodular partial response (nPR), PR, or stable disease after completing PCR to a complete response (CR) after 6 cycles of consolidation with lenalidomide.
* To assess the proportion of patients who convert from a CR with detectable minimal residual disease (MRD) after PCR to a CR with MRD negative state after 6 courses of consolidation with lenalidomide.
* To assess the proportion of patients who convert from a CR with detectable MRD, nPR, PR, or stable disease with residual disease after PCR to a CR with MRD negative state after 6 cycles of consolidation with lenalidomide.
* To monitor and assess toxicity of this regimen.
* To determine if molecular prognostic parameters (e.g., ZAP-70, CD38, cytogenetic abnormalities identified by FISH, IgVH mutation status) relate to response to PCR-lenalidomide therapy.
* To use evaluation of MRD to determine the duration of lenalidomide therapy.
* To determine the progression-free survival in CLL patients using this treatment regimen.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive rituximab IV over 4 hours on days 1 and 2 of course 1, and over 1 hour on day 1 of each subsequent course. Patients also receive pentostatin IV over 30 minutes and cyclophosphamide IV over 30 minutes on day 1, and pegfilgrastim subcutaneously on day 2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Consolidation therapy: Beginning 2 months after completion of induction therapy, patients receive oral lenalidomide once daily on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Continuation therapy: Patients with residual disease continue to receive lenalidomide as in consolidation therapy until they achieve a minimal residual disease-negative status or complete remission. Patients who achieve complete response with no detectable disease discontinue therapy and enter the observation phase.

Blood samples are collected periodically during treatment for translational and pharmacologic studies. Samples are analyzed for immunoglobulin heavy chain gene mutational status, ZAP-70 status, and levels of VEGF, bFGF, thrombospondin, and TGF-beta by ELISA; and for the effects of therapy on immune function. Samples are also stored for future research. Bone marrow aspirate samples are analyzed for minimal residual disease by flow cytometry.

After completion of study treatment, patients are followed every 90 days for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), meeting the following criteria:

  * Biopsy-proven SLL according to WHO criteria
  * CLL diagnosis* according to NCI working group criteria as evidenced by all of the following:

    * Peripheral blood lymphocyte count of > 5,000/mm³
    * Small to moderate peripheral blood lymphocyte with < 55% prolymphocytes
    * Immunophenotyping consistent with CLL defined as:

      * B-cell markers with CD5 antigen in the absence of other pan-T-cell markers (e.g., CD3, CD2)
      * CD19, CD20, or CD23
      * Dim surface immunoglobulin expression
      * Exclusively kappa or lambda light chains
    * Diagnosis of mantle cell lymphoma must be excluded by negative FISH analysis for t(11;14)(IgH/CCND1) on peripheral blood or tissue biopsy or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy NOTE: *Splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
* Previously untreated disease and meets ≥ 1 of the following criteria*:

  * At least 1 or more of the following disease-related symptoms:

    * Weight loss > 10% within the previous 6 months
    * Extreme fatigue attributed to CLL
    * Fevers > 100.5º F for 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure as manifested by the development of or worsening anemia (i.e., hemoglobin ≤ 11 g/dL) and/or thrombocytopenia (i.e., platelet count ≤ 100,000/mm³) not due to autoimmune disease
  * Symptomatic or progressive lymphadenopathy, splenomegaly, or hepatomegaly
  * Progressive lymphocytosis due to CLL with an increase of > 50% over a 2-month period or an anticipated doubling time < 6 months NOTE: *Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease are not sufficient for protocol therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 3.0 times ULN (unless due to Gilbert disease)

  * Direct bilirubin < 1.5 mg/dL for Gilbert disease to be diagnosed if total bilirubin > 3.0 times ULN
* AST and ALT ≤ 3.0 times ULN (unless due to hemolysis or CLL)
* Willing to provide blood samples
* Able to take acetylsalicylic acid (ASA) (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use low molecular weight heparin)
* Not pregnant or nursing
* Negative pregnancy test
* Female patients must use effective double-method contraception beginning 1 month prior to, during, and for 4 weeks after completion of study treatment
* Male patients must use effective contraception during and for 4 weeks after completion of study treatment
* No comorbid conditions, including any of the following:

  * New York Heart Association class III or IV heart disease
  * Recent myocardial infarction (< 1 month)
  * Uncontrolled infection
  * Infection with HIV/AIDS
* No other active primary malignancy requiring treatment or that limits survival to ≤ 2 years
* No history of deep venous thrombosis or pulmonary embolism ≤ 12 months prior to study registration
* No active hemolytic anemia requiring immunosuppressive or other pharmacologic therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or monoclonal antibody-based therapy for treatment of CLL
* Nutraceutical treatments with no established benefit in CLL (e.g., epigallocatechin gallate or other herbal treatments) are not considered prior therapy
* More than 4 weeks since prior radiotherapy
* At least 4 weeks since prior major surgery
* No concurrent corticosteroids

  * Concurrent low doses of steroids (e.g., < 10 mg of prednisone or equivalent dose of other steroid) used for treatment of non-hematologic medical conditions allowed
  * Prior use of corticosteroids allowed
* No prior thalidomide or lenalidomide
* No concurrent therapeutic doses of coumadin-derivative anticoagulants (e.g., warfarin)

  * Doses of ≤ 2 mg daily allowed for thrombosis prophylaxis
  * Prophylactic doses of low molecular weight heparin allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tait D. Shanafelt, MD, Study Chair — Mayo Clinic; Han Win Tun, MD, Principal Investigator — Mayo Clinic; Jose F. Leis, MD, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five (45) participants were recruited at Mayo Clinic (Rochester, Florida and Arizona) between March 2009 and December 2009.
Pre-assignment Details: One participant was deemed ineligible and is excluded from all analyses per study design.
Period: Overall Study
Arm/Group | PCR-Lenalidomide
Started | 44
Completed | 39
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | PCR-Lenalidomide
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 44
Fluorescence In Situ Hybridization (FISH) Abnormalities [Number; unit: participants] — This test determines the presence of abnormalities in specific chromosomes of CLL cells, which are associated with more or less aggressive forms of cancer. Patients with abnormalities of chromosome 11 (deletion 11q23) and 17 (deletion 17p13) experience rapid progression of their CLL.
  participants
    deletion(13q14.2) | 13
    Trisomy 12 | 7
    deletion (11q22) | 6
    17p- | 1
    Other | 2
    Normal | 15
Rai Stage [Number; unit: participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL); higher stages reflect increasing severity.> Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis and lymphadenopathy, Rai Stage II: Lymphocytosis and hepatomegaly +/- splenomegaly, Rai Stage III: Lymphocytosis and anemia, Rai Stage IV: Lymphocytosis and thrombocytopenia
  participants
    Stage I-II | 27
    Stage III-IV | 17
ZAP-70 Status [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive ZAP-70 (>=20%) tend to experience a more aggressive course of CLL.
  participants
    Positive (>=20%) | 24
    Negative (<20%) | 20
CD38 Status [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive CD38 (>=30%) tend to experience a more aggressive course of CLL.
  participants
    Positive (>=30%) | 14
    Negative (<30%) | 30
Immunoglobulin Variable Heavy Chain (IGVH) Mutation Status [Number; unit: participants] — IGVH testing helps predict which patients will experience a more aggressive (if the gene is unmutated, <=2%) or less aggressive (if the gene is mutated, >2%) course of CLL. This technically complex test is only available at select medical institutions.
  participants
    Unmutated | 22
    Mutated | 20
    Not tested | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: A complete response, as defined by the National Cancer Institute Working Group (NCIWG), requires all of the following for a period of at least 2 months:
  - CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PCR-Lenalidomide
Number analyzed (Participants) | 44
participants | 14

2. Secondary Outcome: Number of Participants Who Convert From a Nodular Partial Response (nPR), Partial Response (PR), or Stable Disease (SD) After Pentostatin, Cyclophosphamide, and Rituximab (PCR) to a Complete Response (CR) After 6 Courses of Consolidation With Lenalidomide
Description: According to the NCIWG criteria, response is defined as follows:
  nPR: Meets all criteria for CR, as described above, except the presence of residual clonal nodules in the bone marrow PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100000/μL platelets, >11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions SD: participant who does not meet any of the criteria described above
Time Frame: 12 months
Population: All patients that began lenalidomide consolidation with either and nPR, PR, or SD were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PCR-Lenalidomide
Number analyzed (Participants) | 21
Participants | 5

3. Secondary Outcome: Number of Participants Who Convert From a CR With Minimal Residual Disease (MRD) Positive Status After PCR to a CR With MRD-negative Status After 6 Courses of Consolidation With Lenalidomide
Description: MRD refers to small number of leukemic cells that remain in the participant during treatment or after treatment when the participant has achieved CR. For all participants who achieved CR, the follow-up bone marrow sample was tested for malignant B cells to determine if there was any MRD.
Time Frame: 12 months
Population: All patients that began consolidation with a CR and MRD-negative status were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PCR-Lenalidomide
Number analyzed (Participants) | 5
Participants | 4

4. Secondary Outcome: Number of Participants With a Response (CR, nPR, PR)
Description: Response criteria described in above outcomes.
Time Frame: During treatment (up to 5 years)
Population: All patients that registered to this trial with the intent-to-treat were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PCR-Lenalidomide
Number analyzed (Participants) | 44
Participants | 38

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from registration to death of any cause. Participants were followed for a maximum of 5 years from registration. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: time from registration to death (up to 5 years)
Population: All patients who registered were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PCR-Lenalidomide
Number analyzed (Participants) | 44
months | NA [NA to NA] — Too few events took place during treatment and follow up to obtain a median value and estimate the 95% CI.

6. Secondary Outcome: Treatment Free Survival (TFS)
Description: Treatment Free Survival (TFS) was defined as the time from registration to the earliest date documentation of subsequent treatment or death, whichever came first. Participants were followed for a maximum of 5 years from registration. The median TFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: time from registration to progression (up to 5 years)
Population: All patients that registered to treatment were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PCR-Lenalidomide
Number analyzed (Participants) | 44
months | NA [48 to NA] — Too few events occurred to obtain a median or upper bound of the 95% CI.

ADVERSE EVENTS:
Arm/Group | PCR-Lenalidomide
Serious Adverse Events (participants affected / at risk) | 9/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCR-Lenalidomide (N=44)
Atrial flutter (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper airway infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6)
Platelet count decreased (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCR-Lenalidomide (N=44)
Anemia (Blood and lymphatic system disorders) | 40 (231)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (4)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (11)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8)
Chills (General disorders) | 4 (4)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 28 (116)
Fever (General disorders) | 20 (26)
Pain-Chest (General disorders) | 1 (1)
Syndromes (General disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 3 (3)
Abdominal infection (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Blood Infection (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (2)
Lymph gland infection (Infections and infestations) | 1 (1)
Lymphatic infection (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 4 (4)
Sinus infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin (cellulites) infection (Infections and infestations) | 1 (1)
Upper airway infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin (Investigations) | 1 (1)
Leukopenia (Investigations) | 34 (227)
Neutrophil count decreased (Investigations) | 38 (231)
Platelet count decreased (Investigations) | 32 (262)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 25 (48)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes